CLINICAL TRIAL: NCT06780813
Title: Supplemental Administration of High Flow Oxygen to Enhance Postoperative Recovery and Reduce Infections in Obese Gynecological Cancer Patients
Brief Title: Supplemental High Flow Oxygen to Reduce Infections in Obese Gynecological Cancer Patients
Acronym: SAFE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National and Kapodistrian University of Athens (Other)
Responsible Party: Principal Investigator, Vasilios Pergialiotis, Assistant Professor, National and Kapodistrian University of Athens
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 834/24
Record Dates: First submitted 2025-01-09; First posted 2025-01-17 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Supplemental Oxygen; Gynecological Cancer; Surgical Site Infections
Keywords: Supplemental oxygen; Surgical site infections; Gynecological cancer
MeSH Terms: conditions — Surgical Wound Infection | interventions — Oxygen

STUDY DESIGN:
Intervention Model Description: Patients will be assigned with computer-generated randomization in two groups: i) the group receiving supplemental oxygen in the form of a Venturi mask upon low oxygen saturation in oximetry (SaO2<95%) and a nasal oxygen mask in all other cases during the first 2 postoperative days (phase of hemostasis and inflammation of the surgical wound as well as ii) the control group in which supplemental oxygen will not be administered beyond the basic indications (low saturation, respiratory dysfunction).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supplemental oxygen (Active Comparator): This group will receive supplemental oxygen in the form of a Venturi mask upon low oxygen saturation in oximetry (SaO2<95%) and a nasal oxygen mask (in case of normal oxygen saturation) for the first 2 postoperative days
  Interventions: Behavioral: Supplemental oxygen therapy
- Control group (No Intervention): This group will not receive supplemental oxygen during the first two days of hospitalization

INTERVENTIONS:
Behavioral: Supplemental oxygen therapy — In this grou participants will receive supplemental oxygen in the form of a Venturi mask upon low oxygen saturation in oximetry (SaO2<95%) and a nasal oxygen mask in all other cases during the first 2 postoperative days
  Arms: Supplemental oxygen

SUMMARY:
The incidence of surgical-site infection (SSI) and complications related to wound healing reaches 10-20% of gynecological cancer patients. Each complication may dramatically prolong the hospitalization period and increase the economic burden of hospital care. Appropriate wound care and tissue oxygenation are of special importance for wound healing. Assuming adequate perfusion, the easiest, safest, and most effective way to improve tissue oxygenation is to increase the fraction of inspired oxygen. However, there is considerable controversy as to whether supplemental oxygen actually reduces SSI and healing-related complications as to date, there is absence of relevant data.

DETAILED DESCRIPTION:
This study aims to investigate the prophylactic value of postoperative oxygen administration against the development of wound infections in obese gynecological oncology patients undergoing laparotomy for the treatment of endometrial or ovarian cancer. At the same time, the factors that lead to an increase in this risk will be outlined.

ELIGIBILITY:
Inclusion Criteria:

* Obese (BMI>30kg/m2) gynecological cancer patients
* Optimized preoperative CBC values (hemoglobin >11g/dl, WBC 4.000-11.000 X 109/L, platelets 150,000 to 400,000 X 109/L)
* In the case of neoadjuvant therapy an interval longer than three weeks between the last cycle and the operation

Exclusion Criteria:

* Active immunosuppresion
* Preexisting infection of the abdominal wall
* Preexisting sepsis

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 400 (Estimated)
Dates: Start 2025-01-10 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Surgical site infections | Within 30 days from the operation
  Surgical site infections will be evaluated using the Southampton wound scoring system
Systemic inflammatory response syndrome | Within 30 days from the operation
  The proportion of patients developing SSI-related systemic inflammatory response will be documented

SECONDARY OUTCOMES:
Need for surgical debridement | Within 30 days from the operation
  Need for surgical debridement (bedside or on the operation theatre)
Seroma formation | Within 30 days from the operation
  The development of wound seroma will be recorded
Wound hematoma | Within 30 days from the operation
  The formation of wound hematoma will be evaluated
Uncomplicated wound healing | Within 30 days from the operation
  The proportion of patients with no apparent wound healing problems will be documented
Additional wound assisting devices | Within 30 days from the operation
  The need for vacuum assisted wound healing will be documented
Antibiotic coverage | Within 30 days from the operation
  The need for supplemental antibiotic coverage will be documented
Multidrug resistant pathogens | Within 30 days from the operation
  The proportion of patients with multidrug-resistant pathogens involving SSI will be documented
Duration of hospitalization | Within 30 days from the operation
  The total duration of hospitalization will be documented
Hospital readmissions related to SSI | Within 30 days from the operation
  Readmissions related to SSIs will be documented

OTHER OUTCOMES:
Infectious morbidity | Within 30 days from the operation
  Other infectious morbidity, including urinary tract, pulmonary and gastrointestinal infections will be recorded
Postoperative morbidity | Within 30 days from the operation
  Postoperative morbidity non-related to SSI will be documented using the Clavien-Dindo scaling score
Non-SSI related hospital readmissions | Within 30 days from the operation
  Hospital readmission rates that are not attributed to SSIs will be documented

CONTACTS AND LOCATIONS:
Overall Officials: Nikolaos Thomakos, Associate Professor, Study Director — National and Kapodistrian University of Athens
Locations (1):
- First department of Obstetrics and Gynecology, Athens, Greece

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared for this study